CLINICAL TRIAL: NCT06166979
Title: Assessment of Colonization and Scalp Quality Parameter Improvement by Topical Application of Probiotic Micrococcus Luteus Q24 in Healthy Adults.
Brief Title: Colonisation of Scalp by Topical Probiotic Micrococcus Luteus Q24
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BLIS Technologies Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: BLTCT2023/1
Record Dates: First submitted 2023-12-04; First posted 2023-12-12 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Microbial Colonization
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Intervention Model Description: This is a randomized double-blind baseline controlled pilot study with no crossover.
Who Masked: Investigator
Masking Description: Both participants and investigator are blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study Group A: Probiotic Micrococcus luteus Q24 serum (high dose) (Active Comparator): Group A: Probiotic Micrococcus luteus Q24 serum (dose: 1e8 colony forming units per application)
  Interventions: Other: Active Comparator: Study Group A: Blis Q24 Serum at higher dose
- Study Group B: Probiotic Micrococcus luteus Q24 serum (low dose) (Active Comparator): Group : Probiotic Micrococcus luteus Q24 serum (dose: 1e6 colony forming units per application)
  Interventions: Other: Active Comparator: Study Group B: Blis Q24 Serum at lower dose

INTERVENTIONS:
Other: Active Comparator: Study Group A: Blis Q24 Serum at higher dose — Active Comparator: Study Group A: Blis Q24 Serum at 1e8 cfu/ dose (Active)
  Arms: Study Group A: Probiotic Micrococcus luteus Q24 serum (high dose)
Other: Active Comparator: Study Group B: Blis Q24 Serum at lower dose — Active Comparator: Study Group A: Blis Q24 Serum at 1e6 cfu/ dose (Active)
  Arms: Study Group B: Probiotic Micrococcus luteus Q24 serum (low dose)

SUMMARY:
The purpose of this study is to evaluate the skin quality improvement and colonization efficacy following the application of probiotic Micrococcus luteus Q24 (BLIS Q24) to the scalp from a serum format in healthy adults.

DETAILED DESCRIPTION:
This is a randomized double-blind baseline controlled pilot study with no crossover for the assessment of any changes to the microbial make-up of the skin (The local skin microbiome), detection of colonization by the probiotic bacterium (BLIS Q24) on the skin on the scalp and to evaluate the changes in skin quality parameters following topical application of probiotic in a serum format.

ELIGIBILITY:
Inclusion Criteria:

1. In general, good health, is 18 - 80 years of age.
2. Practice good general body and hair hygiene.

Exclusion Criteria:

1. Have a history of autoimmune disease or are immunocompromised (have a weakened immune system).
2. Free from any scalp disease, active cut, or open wound
3. On hair loss treatment at least 2 months prior to sampling.
4. Have used anti-dandruff shampoos on the scalp and hair for at least 1 week prior to the trial.
5. On concurrent antibiotic or antifungal therapy or regular antibiotic or antifungal. use within the last 1 week.
6. People with allergies or sensitivity to dairy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-02-25 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Change in microbial composition following application of 1e8 cfu per dose Micrococcus luteus Q24 in serum from Day 0 (baseline) to 15 days | 15 days post intervention
  Study will determine the change in microbial composition following the application of 1e8 cfu per dose serum containing Micrococcus luteus Q24 serum to the scalp. The statistical analysis will be carried out to compare the participants skin swab data from baseline to 15 days across one site with a level of significance of p<0.05. Overall colonization based on percentage of population colonized for different interventions will also be analyzed using appropriate statistical analysis software. Analysis will be performed using bacterial genome sequence analysis of the skin swab samples collected.
Change in microbial composition following application of 1e6 cfu per dose Micrococcus luteus Q24 in serum from Day 0 (baseline) to 15 days | 15 days post intervention
  Study will determine the change in microbial composition following the application of 1e6 cfu per dose serum containing Micrococcus luteus Q24 serum to the scalp. The statistical analysis will be carried out to compare the participants skin swab data from baseline to 15 days across one site with a level of significance of p<0.05. Overall colonization based on percentage of population colonized for different interventions will also be analyzed using appropriate statistical analysis software. Analysis will be performed using bacterial genome sequence analysis of the skin swab samples collected.
Change in Skin quality parameters following application of 1e8 cfu per dose Micrococcus luteus Q24 in serum from Day 0 (baseline) to 15 days | 15 days post intervention
  Study will determine the change in skin quality parameters following the application of 1e8 cfu per dose serum containing Micrococcus luteus Q24 serum to the scalp. The statistical analysis will be carried out to compare the participants skin swab data from baseline to 15 days across one site with a level of significance of p<0.05. Overall colonization based on percentage of population colonized for different interventions will also be analyzed using appropriate statistical analysis software. Analysis will be performed using bacterial genome sequence analysis of the skin swab samples collected.
Change in Skin quality parameters following application of 1e6 cfu per dose Micrococcus luteus Q24 in serum from Day 0 (baseline) to 15 days | 15 days post intervention
  Study will determine the change in skin quality parameters following the application of 1e6 cfu per dose serum containing Micrococcus luteus Q24 serum to the scalp. The statistical analysis will be carried out to compare the participants skin swab data from baseline to 15 days across one site with a level of significance of p<0.05. Overall colonization based on percentage of population colonized for different interventions will also be analyzed using appropriate statistical analysis software. Analysis will be performed using bacterial genome sequence analysis of the skin swab samples collected.
Change in microbial composition following application of 1e8 cfu per dose Micrococcus luteus Q24 in serum from Day 0 (baseline) to 29 days | 29 days post intervention
  Study will determine the change in microbial composition following the application of 1e8 cfu per dose serum containing Micrococcus luteus Q24 serum to the scalp. The statistical analysis will be carried out to compare the participants skin swab data from baseline to 29 days across one site with a level of significance of p<0.05. Overall colonization based on percentage of population colonized for different interventions will also be analyzed using appropriate statistical analysis software. Analysis will be performed using bacterial genome sequence analysis of the skin swab samples collected.
Change in Skin quality parameters following application of 1e8 cfu per dose Micrococcus luteus Q24 in serum from Day 0 (baseline) to 29 days | 29 days post intervention
  Study will determine the change in skin quality parameters following the application of 1e8 cfu per dose serum containing Micrococcus luteus Q24 serum to the scalp. The statistical analysis will be carried out to compare the participants skin swab data from baseline to 29 days across one site with a level of significance of p<0.05. Overall colonization based on percentage of population colonized for different interventions will also be analyzed using appropriate statistical analysis software. Analysis will be performed using bacterial genome sequence analysis of the skin swab samples collected.
Change in microbial composition following application of 1e6 cfu per dose Micrococcus luteus Q24 in serum from Day 0 (baseline) to 29 days | 29 days post intervention
  Study will determine the change in microbial composition following the application of 1e6 cfu per dose serum containing Micrococcus luteus Q24 serum to the scalp. The statistical analysis will be carried out to compare the participants skin swab data from baseline to 29 days across one site with a level of significance of p<0.05. Overall colonization based on percentage of population colonized for different interventions will also be analyzed using appropriate statistical analysis software. Analysis will be performed using bacterial genome sequence analysis of the skin swab samples collected.
Change in Skin quality parameters following application of 1e6 cfu per dose Micrococcus luteus Q24 in serum from Day 0 (baseline) to 29 days | 29 days post intervention
  Study will determine the change in skin quality parameters following the application of 1e6 cfu per dose serum containing Micrococcus luteus Q24 serum to the scalp. The statistical analysis will be carried out to compare the participants skin swab data from baseline to 29 days across one site with a level of significance of p<0.05. Overall colonization based on percentage of population colonized for different interventions will also be analyzed using appropriate statistical analysis software. Analysis will be performed using bacterial genome sequence analysis of the skin swab samples collected.
Change in microbial composition post 7 days of last application of 1e8 cfu of Micrococcus luteus Q24 in serum | 7 days post last intervention
  Study will determine the change in microbial composition following the application of 1e8 cfu per dose serum containing Micrococcus luteus Q24 serum to the scalp. The statistical analysis will be carried out to compare the participants skin swab data at Day 36(i.e. post 7 days from last application) across one site with a level of significance of p<0.05. Overall colonization based on percentage of population colonized for different interventions will also be analyzed using appropriate statistical analysis software. Analysis will be performed using bacterial genome sequence analysis of the skin swab samples collected.
Change in microbial composition post 7 days of last application of 1e6 cfu of Micrococcus luteus Q24 in serum | 7 days post last intervention
  Study will determine the change in microbial composition following the application of 1e6 cfu per dose serum containing Micrococcus luteus Q24 serum to the scalp. The statistical analysis will be carried out to compare the participants skin swab data at Day 36(i.e. post 7 days from last application) across one site with a level of significance of p<0.05. Overall colonization based on percentage of population colonized for different interventions will also be analyzed using appropriate statistical analysis software. Analysis will be performed using bacterial genome sequence analysis of the skin swab samples collected.
Change in Skin quality parameters post 7 days of last application of 1e8 cfu of Micrococcus luteus Q24 in serum | 7 days post last intervention
  Study will determine the change in microbial composition following the application of 1e8 cfu per dose serum containing Micrococcus luteus Q24 serum to the scalp. The statistical analysis will be carried out to compare the participants skin swab data at Day 36(i.e. post 7 days from last application) across one site with a level of significance of p<0.05. Overall colonization based on percentage of population colonized for different interventions will also be analyzed using appropriate statistical analysis software. Analysis will be performed using bacterial genome sequence analysis of the skin swab samples collected.
Change in Skin quality parameters post 7 days of last application of 1e6 cfu of Micrococcus luteus Q24 in serum | 7 days post last intervention
  Study will determine the change in microbial composition following the application of 1e6 cfu per dose serum containing Micrococcus luteus Q24 serum to the scalp. The statistical analysis will be carried out to compare the participants skin swab data at Day 36(i.e. post 7 days from last application) across one site with a level of significance of p<0.05. Overall colonization based on percentage of population colonized for different interventions will also be analyzed using appropriate statistical analysis software. Analysis will be performed using bacterial genome sequence analysis of the skin swab samples collected.

CONTACTS AND LOCATIONS:
Locations (1):
- Blis Technologies Ltd, Dunedin, Otago, New Zealand

IPD SHARING:
Plan to Share IPD: Yes
Data and information in the protocol and the clinical study report will be shared to other researchers and/or in publications in due course.
Supporting Information: Study Protocol, CSR
Time Frame: Study report 3 months after completion of the study.
Access Criteria: Summary study report will be shared by the Principal Investigator upon request if not published in public literature.

REFERENCES:
- [Background] Oh J, Byrd AL, Deming C, Conlan S; NISC Comparative Sequencing Program; Kong HH, Segre JA. Biogeography and individuality shape function in the human skin metagenome. Nature. 2014 Oct 2;514(7520):59-64. doi: 10.1038/nature13786. PMID 25279917
- [Background] Bourdichon F, Casaregola S, Farrokh C, Frisvad JC, Gerds ML, Hammes WP, Harnett J, Huys G, Laulund S, Ouwehand A, Powell IB, Prajapati JB, Seto Y, Ter Schure E, Van Boven A, Vankerckhoven V, Zgoda A, Tuijtelaars S, Hansen EB. Food fermentations: microorganisms with technological beneficial use. Int J Food Microbiol. 2012 Mar 15;154(3):87-97. doi: 10.1016/j.ijfoodmicro.2011.12.030. Epub 2011 Dec 31. PMID 22257932
- [Background] van Rensburg JJ, Lin H, Gao X, Toh E, Fortney KR, Ellinger S, Zwickl B, Janowicz DM, Katz BP, Nelson DE, Dong Q, Spinola SM. The Human Skin Microbiome Associates with the Outcome of and Is Influenced by Bacterial Infection. mBio. 2015 Sep 15;6(5):e01315-15. doi: 10.1128/mBio.01315-15. PMID 26374122